CLINICAL TRIAL: NCT01888393
Title: A Phase 1, Open Label Study to Assess the Pharmacokinetics and Safety of Multiple Doses of Lumacaftor in Combination With Ivacaftor in Subjects With Moderate Hepatic Impairment and in Matched Healthy Subjects
Brief Title: Study of Lumacaftor in Combination With Ivacaftor in Subjects With Moderate Hepatic Impairment and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: VX13-809-010
Record Dates: First submitted 2013-06-20; First posted 2013-06-27 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Hepatic Impairment; Healthy
Keywords: pharmacokinetics, hepatic impairment
MeSH Terms: interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Approximately 12 subjects (male and female) with moderate hepatic impairment
  Interventions: Drug: lumacaftor 200 mg q12h + ivacaftor 250 mg q12h
- Group B (Experimental): Approximately 12 healthy subjects (male and female)
  Interventions: Drug: lumacaftor 200 mg q12h + ivacaftor 250 mg q12h

INTERVENTIONS:
Drug: lumacaftor 200 mg q12h + ivacaftor 250 mg q12h

SUMMARY:
This study is designed to evaluate the pharmacokinetics (PK) and safety of multiple doses of lumacaftor in combination with ivacaftor in subjects with moderate hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

Group A: Subjects with Moderate Hepatic Impairment

* Male and female 18 to 65 years of age (inclusive)
* Satisfy the criteria for moderate hepatic impairment defined as a Child Pugh total score of 7 to 9 (Child Pugh Class B) at the Screening Visit
* Willing and able to comply with schedule visits, treatment, laboratory tests, and contraceptive guidelines.

Group B: Healthy subjects

* Male and female 18 to 65 years of age (inclusive)
* Healthy subjects with no clinically relevant abnormalities identified by a detailed medical history, complete physical examination, including blood pressure and pulse rate measurement, standard 12-lead ECG, and clinical laboratory tests
* Willing and able to comply with schedule visits, treatment, laboratory tests, contraceptive guidelines and other study procedures

Exclusion Criteria:

Group A: Subjects with Moderate Hepatic Impairment

* History of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject
* Have fluctuating or rapidly deteriorating hepatic function by history or as indicated by significant variations in or worsening of clinical and/or laboratory signs of hepatic impairment within 6 months before the Screening Visit
* Other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver
* Severe hepatic encephalopathy
* Type 1 diabetes mellitus or evidence of poorly controlled type 2 diabetes
* Hepatocellular carcinoma, HIV, hepatitis B/C
* Significant renal dysfunction
* Solid organ or bone marrow transplantation
* History of regular alcohol consumption, drug abuse or regular smoking

Group B: Healthy subjects

* History of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject
* History of regular alcohol consumption, drug abuse or regular smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Lumacaftor pharmacokinetic parameters, including Cmax, tmax, AUC, Vd, CL/F | 16 days
Ivacaftor pharmacokinetic parameters, including Cmax, tmax, AUC, Vd, CL/F | 16 days

SECONDARY OUTCOMES:
Lumacaftor metabolites pharmacokinetic parameters, including Cmax and AUC | 16 days
Ivacaftor metabolites pharmacokinetic parameters including Cmax, tmax, AUC | 16 days
Safety and tolerability as mentioned by adverse events, clinical laboratory values, standard electrocardiograms, Vital signs and pulse oximetry | 21 days

CONTACTS AND LOCATIONS:
Locations (2):
- Prague, Czechia
- Bratislava, Slovakia